CLINICAL TRIAL: NCT06776822
Title: The Effect of DNS Therapy in Children After Cardiac Surgery
Brief Title: The Effect of DNS Therapy on Asymmetry in Children After Surgery of Congenital Heart Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK-714/24
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease in Children
Keywords: Congenital heart disease; Rehabilitation; Complication of surgical treatment; Postural asymmetry; Maximal expiratory pressure; Minimal expiratory pressure
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with congenital heart disease, 6-18 years (Experimental)
  Interventions: Other: Dynamic neuromuscular stabilisation

INTERVENTIONS:
Other: Dynamic neuromuscular stabilisation — The nervous system establishes programs that control human posture, movement and gait. This 'motor control' is largely established during the first critical years of life. Therefore, the "Prague School" emphasizes neurodevelopmental aspects of motor control in order to assess and restore dysfunction of the locomotor system and associated syndromes.
  Other Names: DNS

SUMMARY:
This thesis will examine the consequences of congenital heart disease (CHD) surgery in children. The main goal of this work is to point out the possible development of late consequences after cardiac surgery in childhood (e.g. asymmetry, scoliosis, hypomobility of the spine) and to assess the effect of DNS therapy on the resolution of the consequences. For patients, after an intensive three-week rehabilitation intervention, an improvement in the monitored initial parameters is expected, which would lead to an improvement in the quality of life.

DETAILED DESCRIPTION:
As part of the diploma thesis, a study will be conducted in patients after cardiac surgery performed at the Motol Hospital within the Children's Cardiology Center. The intervention will be performed in Rehabilitation Clinic Teplice nad Bečvou. The study group will include children aged 6-18 years after VSV surgery without other serious health complications. The subjects will undergo therapy according to DNS for 3 weeks. Therapy according to DNS will take place twice a day (1x individual physiotherapy 40 minutes, 1x group 40 minutes) and will be supplemented with conventional therapy (e.g. scar care).

The initial examination will be performed by a doctor and a trained physiotherapist in a blinded mode (information about which patients are undergoing the intervention will not be known). The initial examination will include imaging of the spine, ideally EOS (low radiation exposure). During the initial and final examination, a trunk stabilization examination will be performed according to the DNS protocol with photo documentation, the values of MIP and MEP oral pressures (cm H₂O) will be measured, the symmetry index will be measured using the SCODIAC software, the mobility of the spine will be examined (Schober distance, Stibor distance, Otto inclination distance, Thomayer distance, in cm) and the respiratory amplitudes on the chest will be measured (mesosternal and xiphosternal, in cm). The subjects will complete the SF-36 quality of life questionnaire before the start of therapy and after its completion. The parameters will be compared during the initial and final examination.

ELIGIBILITY:
Inclusion Criteria:

* children 6-18 years, surgery of congenital heart disease

Exclusion Criteria:

* any other disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mobility of the spine - Stibor distance | From enrollment to the end of treatment at 3 weeks
  The Stibor distance shows the development of the thoracic and lumbar spine. The starting point is the spine of the L5 vertebra, the second point is the spine of the C7 vertebra. The distance between them is measured and its change during relaxed forward bending are observed. A healthy spine should lengthen by 7-10 cm.
Mobility of the spine - Otto's inclination distance | From enrollment to the end of treatment at 3 weeks
  Otto's inclination distance measures the mobility of the thoracic spine during forward bending. The starting point is the spine of the C7 vertebra, from which we measure 30 cm caudally. The distance of the points shown increases by at least 3.5 cm with forward tilt.

SECONDARY OUTCOMES:
Maximal and minimal expiratory pressure | From enrollment to the end of treatment at 3 weeks
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) are global measures of maximal strength of respiratory muscles and they are the greater pressure which may be generated during maximal inspiration and expiration against an occluded airway. MEP and MIP are assessed by using a pressure reading device (manometer) and is used for respiratory muscle strength testing to obtain objective measurements of positive (expiratory) and negative (inspiratory) pressures.
Anterior trunk symmetry index (ATSI) | From enrollment to the end of treatment at 3 weeks
  Spinal deformities and postural disorders can be assessed by evaluation of trunk surface deformity. On patients, the anatomical landmarks are highlighted and examined with digital photography of the trunk, taken from the front. After that, the anatomical points are indicated on a digital photo and the index is measured. Pathologic is index above 27. Higher numbers mean more asymmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Safarova, PhD., PhDr., Study Director — Rehabilitation and Sports Medicine Clinic
Locations (1):
- Motol University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Unending - Beginning after publication with no end date
Access Criteria: For anybody interested, the results of the study, on-line